CLINICAL TRIAL: NCT06316596
Title: Evaluation Of Newborn Cerebral Oksigenation With Near Infrared Spectroscopy (NIRS) In Cesarean Section Surgeries Performed With Neuroaksial Blocks
Brief Title: Brain Oxygenation in Newborns Due to Neuroaksial Methods
Acronym: oxygenation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ahsen Gur Celik, Doctor of anesthesiology and reanimation, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2011-KAEK-25 2023/09-16
Record Dates: First submitted 2023-11-17; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Cesarean Section; Pregnancy Related; Cerebral Hypoxia; Anesthesia, Regional; Oxygen Saturation
Keywords: Anesthesia, Spinal; Anesthesia, Epidural; Newborn; Oxygen; Hypotension
MeSH Terms: conditions — Hypoxia, Brain; Hypotension | interventions — Anesthesia, Spinal; Anesthesia, Epidural

STUDY DESIGN:
Intervention Model Description: The research is a prospective controlled,randomized,double-blind study
Who Masked: Participant
Masking Description: The research is a prospective, randomized, single-blind, parallel group study. In the study, the Quincke needle will be used for spinal anesthesia and the Tuoghy needle will be used for epidural anesthesia. Oxygenation will be evaluated with the help of NIRS probe in the post-cesarean newborns of pregnant women who will undergo elective cesarean section.
  Vitals will be monitored throughout the case with electrocardiography (ECG), non-invasive blood pressure monitoring and spO2. The amount of vasopressor agent and hydration required by the mother throughout the case will be recorded. While one anesthesiologist will monitor the anesthesia method and maternal vitals, the other anesthetist will monitor the NIRS monitoring attached to the newborn.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEWBORN BORN AFTER EPIDURAL ANESTHESIA (Active Comparator): Group epidural, 0.5% buvasin® will be applied epidural space in the lateral position after monitoring. The patient will be placed in the supine position and surgery will begin when the T5 spinal level is achieved. Pregnant heart rate, blood pressure and saturation values will be recorded at intervals and iv ephedrine will be administered when there is a 25% or more drop in blood pressure. When there is a 25% or more decrease in heart rate, iv atropine will be administered. A NIRS probe (infant,saturation sensor, Invos , Tullamore, Ireland) and pulse will be attached to the newborn by another anesthetist and the measurements will be recorded. Blood pressure will be taken from the umbilical vein. APGAR(activity,pulse,grimace,appearance,respiration), heart rate, SpO2 and umbilical vein saturation values of the newborn will be recorded. NIRS and spO2 values of the newborn will be checked intermittently.
  Interventions: Procedure: Epidural Anesthesia
- NEWBORN BORN AFTER SPINAL ANESTHESIA (Active Comparator): Group spinal, 0.5% buvasin® heavy will be applied spinal space in the lateral position after monitoring. Surgery will begin when the patient is placed in the supine position and T5 spinal level is achieved. Pregnant heart rate, blood pressure, and saturation values are recorded at regular intervals, and when there is a 25% or more drop in blood pressure, the patient will be given iv ephedrine. When there is a 25% or more drop in heart rate, iv atropine will be administered. A NIRS probe (infant,saturation sensor, Invos , Tullamore, Ireland) and pulse will be attached to the newborn by another anesthetist and the measurements will be recorded. Blood pressure will be taken from the umbilical vein. The newborn's APGAR(activity,pulse,grimace,appearance,respiration), heart rate, SpO2 and umbilical venous saturation values will be recorded. NIRS and spO2 values will be checked intermittently.
  Interventions: Procedure: Spinal Anesthesia

INTERVENTIONS:
Procedure: Spinal Anesthesia — Near infrared spectroscopy , neonatal peripheral oxygen saturation measurements and hemodynamic data will be compared between groups
  Arms: NEWBORN BORN AFTER SPINAL ANESTHESIA
Procedure: Epidural Anesthesia — Near infrared spectroscopy , neonatal peripheral oxygen saturation measurements and hemodynamic data will be compared between groups
  Arms: NEWBORN BORN AFTER EPIDURAL ANESTHESIA

SUMMARY:
Epidural and spinal anesthesia techniques are frequently used all over the world in elective cesarean section operations. To evaluate the effects of epidural and spinal anesthesia techniques applied in cesarean section surgery on neonatal cerebral oxygenation using Near Infrared Spectroscopy (NIRS).

DETAILED DESCRIPTION:
In all newborns, cerebral oxygen goes through a complex process as it moves from the fetus to the newborn stage. The type of delivery, anesthesia management, maternal factors before and during birth, and fetal malformations vary in the time it takes for arterial oxygen saturation to reach the expected level in the transition from the fetus to the newborn stage. NIRS is a regional oxygenation monitoring technique and measures regional oxygen saturation. NIRS can also be used as a non-invasive monitoring technique for cerebral oxygenation and hemodynamics. The transparency of tissue to infrared light (spectrum 700-1000 nm) and the formation of oxygenated hemoglobin (O2Hb) and deoxygenated hemoglobin in cerebral blood vessels within the infrared light.

It is based on absorption by (HHb). Hypotension due to sympathetic system blockade is a common finding in neuraxial blocks. Preventing hypotension in pregnancy and prompt intervention when it develops are important to prevent fetal complications. Determining the best neuraxial method in terms of hemodynamics will guide clinicians in practical use. 80 pregnant women between the ages of 18-35 who are scheduled for cesarean section and newborns after cesarean section will be included in the study. Study randomization will be done in sealed envelopes using computer generated randomization codes by a doctor who will not be involved in newborn baby care. For the quality and standardization of the block, it will be performed by an anesthesiologist experienced in spinal and epidural anesthesia. Pregnant heart rate, blood pressure, and saturation values are recorded at regular intervals, and when there is a 25% or more decrease in blood pressure compared to the initial value, iv ephedrine will be administered to the patient. If the heart rate is 25% and In case of a fall on the baby, iv atropine will be administered. After birth, the newborn will be placed in a pre-heated radiant warmer and normal newborn care will be provided by the newborn team, as is done routinely. A NIRS probe and a right-hand transcutaneous pulse oximeter (spO2) will be attached to the left and right frontal regions of the newborn by another anesthetist (anesthesia technique: blind) participating in the study, other than the person performing the neuraxial block, and the measurements will be recorded by the same person.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18-35 and newborns after cesarean section
* Newborns born >37 weeks of gestation
* ASA II pregnant women

Exclusion Criteria:

* Previous local anesthetic allergy
* Those with bleeding diathesis disorder
* Having a mental disorder
* Those who are allergic to the drugs used
* Patients who did not consent to participate in the study
* Height <1.55 meters. or >1.70 meters.
* Presence of infection in the block area
* Body mass index >35 kg/m²
* Those with gestational hypertension and SAP>140 mmHg or DAP>90 mmHg in three pre-pregnancy measurements
* Known presence of fetal anomaly
* Those with known placenta pathology
* Those with a history of fetal anomaly and abnormal birth in previous pregnancies

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women between the ages of 18-35 and newborns after cesarean section
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Near İnfrared Spectroscopi | on 10 minutes
  Near Infrared Spectroscopy (NIRS,infant,saturation sensor, Invos , Tullamore, Ireland) monitors hemodynamic activity in the brain, offering the potential for cerebral monitoring in the region of interest.NIRS is a probe-guided device used for brain oxygenation in newborns.

SECONDARY OUTCOMES:
Maternal mean arterial pressure | during cesarean section
  Maternal mean arterial pressure is monitored by non-invasive blood pressure measurement
Newborn vitalty | 10 minutes after birth
  Newborn saturation are monitored with peripheral oxygen saturation(spo2,saturation sensor, Drager, Lübeck, Germany)
Newborn vitalty | 10 minutes after birth
  Newborn heart rate are monitored with pulse oximeter(heart rate sensor, Covidien, Dublin, Ireland

CONTACTS AND LOCATIONS:
Overall Officials: Ahsen Gür Çelik, Principal Investigator — gurahsen@gmail.com

IPD SHARING:
Plan to Share IPD: No